CLINICAL TRIAL: NCT03202446
Title: Phase 3 Randomized Clinical Trial Evaluating the Use of the Laser-Assisted Immunotherapy (LIT) System in Advanced Breast Cancer
Brief Title: Randomized Clinical Trial Evaluating the Use of the Laser-Assisted Immunotherapy (LIT/inCVAX) in Advanced Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Eske Corporation S.A.C (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IP-LIT-P003
Record Dates: First submitted 2017-06-16; First posted 2017-06-28 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer Stage IIIA; Breast Cancer, Stage IIIB; Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — glycated chitosan; Cyclophosphamide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: LIT and Placebo (Experimental): Patients receive laser-assisted immunotherapy along with Placebo cyclophosphamide tablets. Patients' laser-assisted immunotherapy treatment will be based on the number and size of laser-accessible solid tumors available at the time of treatment. In and around each photothermal laser-treated site will be injected 1 mL of 1% Glycated Chitosan (GC) Injection, with a total of up to 4 sites being treated per patient. The maximum dose of GC Injection that a patient can receive in 1 visit is 4 mL.
  Interventions: Drug: 1% Glycated Chitosan; Device: Photothermal Laser; Drug: Placebo
- Arm 2: LIT and low-dose Cyclophosphamide (Experimental): Patients will receive laser-assisted immunotherapy and low-dose cyclophosphamide (300 mg, administered orally once per week between treatment weeks 0-11 in each treatment cycle). Patients' laser-assisted immunotherapy treatment will be based on the number and size of laser-accessible solid tumors available at the time of treatment. In and around each photothermal laser-treated site will be injected 1 mL of 1% Glycated Chitosan (GC) Injection, with a total of up to 4 sites being treated per patient. The maximum dose of GC Injection that a patient can receive in 1 visit is 4 mL.
  Interventions: Drug: 1% Glycated Chitosan; Device: Photothermal Laser; Drug: Cyclophosphamide
- Arm 3: Control Arm (Active Comparator): Patients will receive the standard of care.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: 1% Glycated Chitosan
  Other Names: GC
  Arms: Arm 1: LIT and Placebo; Arm 2: LIT and low-dose Cyclophosphamide
Device: Photothermal Laser
  Arms: Arm 1: LIT and Placebo; Arm 2: LIT and low-dose Cyclophosphamide
Drug: Placebo
  Arms: Arm 1: LIT and Placebo
Drug: Cyclophosphamide
  Arms: Arm 2: LIT and low-dose Cyclophosphamide
Drug: Standard of Care
  Arms: Arm 3: Control Arm

SUMMARY:
Our study evaluates the use of Laser-Assisted Immunotherapy (LIT) plus placebo and LIT plus low-dose cyclophosphamide versus that of Standard of Care in patients presenting with Stage IIIA, IIIB or IV breast cancer.

One-third of enrolled patients will receive LIT plus placebo, one-third will receive LIT plus low-dose cyclophosphamide, and one-third will be assigned to a control group that receives Standard of Care.

DETAILED DESCRIPTION:
Laser-Assisted Immunotherapy (LIT) is intended to a systemic anti-tumor immune response by priming a tumor with laser energy to liberate an array of tumor antigens from whole cells, immediately followed by administration of the immune stimulant Glycated Chitosan (GC), which is designed to activate antigen presenting cells and facilitate the uptake of tumor antigens. In turn, the antigen presenting cells activate the patient's immune system, resulting in an immune response towards the remaining tumor(s).

In this study it is investigated if the addition of low-dose cyclophosphamide increases the anti-tumor immune response of LIT, as well as comparing the effect of LIT plus Placebo or LIT plus low-dose cyclophosphamide to a control arm of patients receiving Standard of Care therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age
2. Patient must have measurable disease that has progressed despite their current and past treatment plans and with not more treatments lines available according NCI guidelines, described in the subject medical report.
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Patient has adequate organ function, confirmed by the following laboratory values obtained ≥14 days prior to the first treatment:

   * Bone Marrow Function:

     1. Absolute neutrophil count (ANC) ≥1.5 × 103/mm3
     2. Platelets >75 × 103/mm3
     3. Hemoglobin ≥9 g/dL
   * Hepatic Function:

     1. AST and ALT ≤3 × upper limit of normal (ULN); if liver metastases, then ≤5 × ULN.
     2. Bilirubin ≤2.0 × ULN.
   * Renal Function:

     1. Serum creatinine ≤2.0 × ULN or a creatinine clearance of >60 mL/min the calculation of the creatinine clearance will be performed using the cockcroft gault equation (CRCL).
5. Patient is willing to provide written informed consent and agrees to comply with visit schedule.
6. Patient is willing to participate in yearly follow-up calls for an additional 4 years after the completion of the 12 month study period.
7. Patient has life expectancy ≥ 6 months.
8. Patient has Stage 3b, 3c or stage 4 breast cancer and has a laser-accessible solid tumor that is palpable to touch allowing insertion of interstitial laser fiber without imaging techniques. At least one palpable tumor must be >1 cm with previous treatment failed (no more lines available for patient treatments including chemotherapy, radiation therapy , monoclonal antibodies), described by NCI guidelines and described in the patient's medical report.
9. Patient with relapsed or refractory laser-accessible breast cancer, and where the investigator believes that the patient will not require surgical intervention for at least 12 weeks.
10. Patients who are of child-bearing potential (males and females) using an effective method of contraception during the treatment period and for at least 6 months after the last dose of treatment and patients who are not of child-bearing potential (males and females, e.g.post menopause). Women of child-bearing potential must have a negative serum pregnancy test just prior to first treatment. The study will provide a barrier method (e.g. condoms, etc).
11. Patient fits into the pre-defined stratification schedule

Exclusion Criteria:

1. Patient has received prior treatment with glycated chitosan or laser-assisted immunotherapy GC Injection.
2. Patient has a known allergic reaction to shellfish, crabs, crustaceans, or any study components used in treatment.
3. Patient has symptomatic or untreated CNS disease, including seizures. Patients with asymptomatic CNS metastases are eligible provided that they have been clinically stable for a minimum of 4 weeks and are not on steroid treatment.
4. Patient has impaired cardiac function of clinical significance or has experienced within 6 months of initiation of treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
5. Patient has an implantable pacemaker or cardioverted defibrillator within 5 cm of the laser-accessible solid tumor to be treated with laser-assisted immunotherapy.
6. Patient has uncontrolled hypertension.
7. Patient has an ongoing requirement for therapeutic anticoagulation therapy (low-dose anticoagulants or low molecular weight heparin for the prevention of deep vein thrombosis and maintenance of patency of central venous devices is allowed)
8. Patient has HIV or AIDS or history of chronic hepatitis B or C (those who are considered cured of chronic hepatitis B or C may be allowed). Physician may test the patient for hepatitis and exclude the patient if the test is positive.
9. Patient has a serious autoimmune disease (e.g., Lupus). Consultation with medical monitor is required to discuss enrollment if patient has autoimmune disease.
10. Patient has an active infection requiring antibiotics.
11. Patient has presence of ascites or pleural effusion requiring chronic medical intervention.
12. Patient is receiving concomitant treatment with systemic corticosteroids (e.g., predisone) or other immunosuppressive therapy (e.g., methotrexate). Patient should be free of corticosteroid use for at least 18 weeks prior to trial enrollment
13. Patient has received treatment with chemotherapy, radiation, hormones, antibody or other immunotherapy, gene therapy, vaccine therapy, or an investigational product like a treatment for cancer within 4 weeks prior to the start of the study treatment or within 5 t1/2 of a drug, whichever is shorter.
14. Patient has unresolved toxicities from prior anticancer therapy that may limit the ability to remain in the study.
15. Patient has had a surgical procedure ≤14 days prior to the first scheduled treatment; in all cases, the patient must be sufficiently recovered and stable before treatment administration.
16. Patient has any serious or unstable concomitant systemic conditions that are incompatible with this clinical study (e.g., substance addiction, psychiatric disturbance, or uncontrolled intercurrent illness including active infection, arterial thrombosis, abnormal hyper-coagulation profile, or symptomatic pulmonary embolism) or would complicate the study.
17. Patient has any other condition that may cause an increased risk associated with the study participation or may interfere with the interpretation of study results, and in the opinion of the investigator, would make the patient inappropriate for entry into this study.
18. Patient is pregnant, lactating, or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Assessed as week 52
  Overall response rate (ORR) (defined as the percent of patients within each treatment group that achieved complete or partial response, according to irRC, at the end of week 52) comparison between each LIT group and control group.

SECONDARY OUTCOMES:
Overall Survival | Week 0 through Week 52 of study period
  Overall survival (OS): There will be an OS comparison between the treatment arms 1 and 2 vs. control arm at the end of the 52 week trial.
Relative change in overall tumor burden | Week 0 through Week 52 of study period
  Patients demonstrate a 20% improved relative overall change of total tumor burden compared to the control group at the end of the 52 week trial period.
Health Related Quality of Life (HRQOL) | Week 0 through Week 52 of study period
  To assess and compare the HRQOL of those that receive laser-assisted immunotherapy vs Control. HRQOL refere to a multidimensional assessment that includes at least the physical, emotional (or psychological) and social domain, and may also include cognitive functioning, sexuality, and spirituality. The Assessment will be QOL Scale/Breast Cancer designed by NATIONAL MEDICAL CENTER AND BECKMAN RESEARCH INSTITUTE.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Freitas, MD, Principal Investigator — Ricardo Palma Clinica
Locations (4):
- Peru (4):
  - Clinica Ricardo Palma, Lima
  - Hospital Maria Auxiliadora, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima

IPD SHARING:
Plan to Share IPD: Undecided